CLINICAL TRIAL: NCT05640557
Title: The Effect of an Exercise Program Designed for Young Instrumentalists (Musicians) on Music Performance Anxiety
Brief Title: Exercises and Performance Anxiety Among Young Instrumentalists.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anna Cygańska (Other)
Responsible Party: Sponsor-Investigator, Anna Cygańska, Principal Investigator, PhD in physical culture science, Józef Piłsudski University of Physical Education
Organization: Józef Piłsudski University of Physical Education (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SKE 01-26/2022
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Musculoskeletal Pain; Performance Anxiety
Keywords: Occupational Stress; Musculoskeletal Pain; Performance anxiety; Occupational Diseases; Exercise Therapy
MeSH Terms: conditions — Musculoskeletal Pain; Occupational Stress; Occupational Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There will be two groups: study group (taking a part in the exercise program) and control (no intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The participants of the study will take part in exercises (proprietary exercise program), 2 times per week, 45 minutes, for 6 weeks. They will be measured before and after the 6-week exercise program.
  Interventions: Other: Physical Exercises
- Control group (No Intervention): The study participants will not be subjected to any intervention, they will be measured twice, 6 weeks apart. They will be asked to lead their habitual lifestyle.

INTERVENTIONS:
Other: Physical Exercises — An original, noninvasive exercise program
  Arms: Experimental group

SUMMARY:
The purpose of this study is to assess the impact of an original exercise program intended for students of the University of Music on dealing with stage fright and its psychophysical symptoms.

DETAILED DESCRIPTION:
The study group covers students of a music university who play various musical instruments. Participants will be divided into the experimental and control groups. The study duration is scheduled to be 6 weeks. The control group will not have any intervention. The experimental group will undertake 45 mins exercise classes twice a week. Each exercise session will consist of an initial part (warm-up), a main part with exercises designed to strengthen the postural muscles and stretch the contracted muscle groups that are especially prone to pain in musicians (back and upper limbs), and a final part of calming and breathing exercises.

At the beginning and at the end of the study, participants of both groups will be asked to complete a Polish version of validated psychological questionnaires: Kenny Music Performance Anxiety Inventory-Revised, Ogińska-Bulik's & Juczyński's Resiliency Assessment Scale (SPP-25), Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians of the Polish Population (MPIIQM-P) and one original questionnaire assessing the stress level before, during and after a performance. All participants will also undergo physical examination. A measurement of the range of motion of trunk flexion in standing (cm) and the algometric measurement of the pain threshold (kg/cm2) of selected back muscles (trapezius muscles, upper and lower and levator scapula) on the right and left sides of the body. Algometric measurements will be made using the Pain Test FPX algometer Algometer (Wagner).

Statistical analysis. The variables will be coded and analyzed using the STATISTICA program. Baseline demographics will be compared between groups (independent t-tests, chi-square tests). Two-way mixed-model analyses of variance (ANOVA) will explore the effect of the exercise program on symptoms and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* playing on a musical instrument for at least 5 years
* age 18 to 35
* consent to participate in the study
* participation in at least 8 meetings (exercise) within 6 weeks

Exclusion Criteria:

* current (last 3 months) locomotor injuries (fractures, sprains, dislocations), medical contraindications to exercise, confirmed by a medical opinion
* neurological and oncological diseases confirmed by a medical diagnosis
* previous spine surgeries, scoliosis confirmed by radiograph (<10ᵒ Cobb)
* regular intake of muscle relaxants, painkillers, anti-inflammatory drugs, anti-depressants
* age under 18 or over 35
* no consent to participate in the study to participate in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety level - total | Before starting the study
  Kenny Music Performance Anxiety Inventory - Certified Polish translation; the total score in the questionnaire shows the strength of stage fright; the higher the score, the greater the stage fright; from 0 to 240;
Anxiety level - specific psychological predispositions (SPP) | Change between Baseline and post-treatment, 6 weeks
  Kenny Music Performance Anxiety Inventory - Certified Polish translation; the higher the score, the worse the specific psychological predispositions; from 0 to 96;
Pain Interference | Change between Baseline and post-treatment, 6 weeks
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P); from 0 to 50, the higher the score, the greater the pain interference;
Pain Intensity | Change between Baseline and post-treatment, 6 weeks
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P); from 0 to 40, the higher the score, the greater the pain intensity;
Anxiety level - biological predisposition (BP) | Change between Baseline and post-treatment, 6 weeks
  Kenny Music Performance Anxiety Inventory - Certified Polish translation; the higher the score, the worse the biological predisposition; from 0 to 30;

SECONDARY OUTCOMES:
Flexibility level | Change between Baseline and post-treatment, 6 weeks
  Trunk flexion assessment in standing in centimeters
Resilience level | Before starting the study
  The Polish Version of the Resilience Scale 25; The higher the score obtained on the scale, the higher it is resilience is presented by the person completing the questionnaire (from 0 to 100; 0-65 - means low resilience, 66-77 - means medium resilience, and 78-100 means high resilience);
Changes in algometric measurements | Change between Baseline and post-treatment, 6 weeks
  The algometric measurement concerns the assessment of muscle pressure sensitivity - pain threshold in kg/cm2 made using the Pain Test FPX Algometer (Wagner).
Anxiety level - general psychological predisposition (GPP) | Before starting the study
  Kenny Music Performance Anxiety Inventory - Certified Polish translation; the higher the score, the worse the general psychological predisposition; from 0 to 114;
Anxiety level during last performance | Change between Baseline and post-treatment, 6 weeks
  Authors own questionnaire; the higher the score, the greater the stage fright; from 5 to 30;
Assessment of exercises an program | After 6 weeks of exercise program
  Authors own questionnaire; the higher the score, the higher the rating of the original exercise program; from16 to 96;

OTHER OUTCOMES:
Age | Before starting the study
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Gender | Before starting the study
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Instrument played | Before starting the study
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Practice time (years) | Before starting the study
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Weekly practice time (hours) | Before starting the study
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Presence of pain | Baseline and after 6 weeks
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Localisation of pain (number) | Baseline and after 6 weeks
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Localisation of pain (body area) | Baseline and after 6 weeks
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)
Prevalence of pain | Baseline and after 6 weeks
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P)

CONTACTS AND LOCATIONS:
Overall Officials: Anna K. Cygańska, Doctor, Principal Investigator — Józef Piłsudski University of Physical Education in Warsaw
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No